CLINICAL TRIAL: NCT06372626
Title: A Phase I/II Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of ZG005 in Combination With Etoposide and Cisplatin in Participants With Advanced Neuroendocrine Carcinoma.
Brief Title: Study of ZG005 in Combination With Etoposide and Cisplatin in Participants With Advanced Neuroendocrine Carcinoma.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZG005-004
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Etoposide; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Dose-escalation study of ZG005 in combination with Etoposide and Cisplatin.
  Interventions: Biological: ZG005; Drug: Etoposide; Drug: Cisplatin
- Part 2: Dose Expansion (Experimental): Group A: ZG005 in combination with Etoposide and Cisplatin; Group B: Placebo in combination with Etoposide and Cisplatin.
  Interventions: Biological: ZG005; Drug: Etoposide; Drug: Cisplatin; Drug: Placebo

INTERVENTIONS:
Biological: ZG005 — ZG005 for dose escalations are set as 10mg/kg, 20mg/kg, and the other doses after discussion. intravenous infusion, once every 3 weeks.
  ZG005 for dose expansion will commence after the Recommended Phase 2 Dose (RP2D) is determined during the dose-escalation stage.
Drug: Etoposide — IV infusion
Drug: Cisplatin — IV infusion
Drug: Placebo — 0.9% Sodium Chloride Injection
  Arms: Part 2: Dose Expansion

SUMMARY:
The trial is divided into two parts. PART 1 is a dose escalation study of the ZG005 combined with Etoposide and Cisplatin, primarily assessing the tolerability and safety of this combined treatment. PART 2 is a dose expansion study, further evaluating the preliminary efficacy and safety of this combined treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Male or female 18-70 years of age.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Histologically confirmed recurrent or metastatic neuroendocrine carcinoma
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Medical history, computed tomography or magnetic resonance imaging results indicate that existence of the central nervous system metastases;
* Any other malignancy within 5 years.
* participants were deemed unsuitable for participating in the study by the investigator for any reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 2 years
Objective Response Rate (ORR) | Up to 2 years
  ORR was defined as the percentage of the participants in the analysis population who have a Complete Response or a Partial Response. The ORR per RECIST 1.1 as assessed by Investigator is presented
Adverse Event (AE) | Up to 2 years
  Number of participants with adverse events that are related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No